CLINICAL TRIAL: NCT04619589
Title: Characterization of Dyschromic Hypertrophic Scar: An Observational Clinical Trial
Brief Title: Characterization of Dyschromic Hypertrophic Scar
Status: Completed | Type: Observational
Sponsor: Medstar Health Research Institute (Other)
Responsible Party: Sponsor
Other Study IDs: Study430
Record Dates: First submitted 2020-11-02; First posted 2020-11-06 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Burn Scar; Hypertrophic Scar; Hyperpigmentation; Hypopigmented Scar
Keywords: burn; scar; hypertrophic scar; dyspigmentation; dyschromic scar
MeSH Terms: conditions — Cicatrix, Hypertrophic; Hyperpigmentation; Burns; Cicatrix

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Skin tissue and blood samples will be obtained. Blood and skin tissue will be coded with unique identifying numbers and maintained in our lab. Samples that are not completely used in this study may (with the permission of the subject via Informed Consent and HIPAA Authorization) be transferred to an existing Biospecimen Repository (MedStar IRB #2012- 233) and stored indefinitely.
  All biologic samples, as well as genomic data, are subject to withdrawal from their respective repositories at any time upon request of the research participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Currently, there are limited prevention or treatments available for dyschromia in burn hypertrophic scars (HTSs). The limited available techniques involve transferring melanocytes from unaffected areas to the scar to adjust pigment. These techniques involve the creation of a donor site and do not utilize the cells that may already be present in scars. This study aims to confirm melanocyte presence in regions of hypo- and hyper- pigmented HTS. If melanocytes can be found in regions of hypopigmentation, these scars may be able to be treated in the future by pigmentation stimulators without the need for surgery. Additionally, if pigmentation specific molecules of interest can be found to be up-regulated in hyperpigmented scar, these may be able to be altered by a pharmacotherapy.

DETAILED DESCRIPTION:
Subjects with burn scars that are lighter and/or darker than their normal skin will be asked to participate in this study. It is being done to obtain more information about why some people develop scars that are different in color to their normal skin after trauma to the skin such as a burn.

Participants who wish to participate will have scar measured with a ruler, and study sites identified and photographed.

Additionally the following procedures will be done:

Non-invasive measurements: Each area of scar will have multiple non-invasive measurements done. These include:

* scar scales - subjective measures of color, itching, pain, height, etc.
* elasticity - a probe is briefly placed on top of the skin to measure its ability to stretch
* induration - a probe is briefly placed on top of the skin to measure how firm it is
* color - a skin probe in briefly placed on top of the skin to measure its color

Biopsies: Based on the measurement of the scars, several small 3mm punch biopsies will be done. Subjects with light colored scars and total scar greater than 500cm2 are eligible to participate in an optional sub-study. For this sub-study, an additional excisional biopsy 1 cm by 2 cm in the shape of an oval will be obtained from the lighter colored scar.

Blood collection: Blood will be collected for correlating blood characteristics to scar outcome. Approximately 20 mL of blood will be collected, which is less than 2 tablespoons. A portion of this blood might be used in the future for genome sequencing of pigmentation or hypertrophic scar-related gene sequences. Whole genome sequencing will not be performed.

Interview: Personal information, medical history, health behaviors, and scar history will be reviewed.

Data collection: Information about initial burn injury, hospitalization, and outpatient visits will be requested from the medical record.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age or older
* Skin trauma resulting in a dyschromic scar

Exclusion Criteria:

* Dyschromic scar dole to face, genitals, fingers, or toes
* Known Lidocaine allergy
* Pregnancy
* Prisoner Status

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects eligible for this study will have a dyschromic scar following thermal, chemical, or electrical trauma.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2023-06-28 (Actual); Study Completion 2023-06-28 (Actual)

PRIMARY OUTCOMES:
Identify Melanocyte Presence | 1 year
  Confirm melanocyte presence in regions of hyper- and hypo-pigmented HTS, as well as normal skin by multiple assays including en face staining and immunofluorescent staining with melanocytes markers.

SECONDARY OUTCOMES:
Characterize Pigmentation Signaling | 1 year
  Compare pigmentation signaling molecules between hyper-, hypo-, and normally pigmented scar and skin using immunofluorescent staining and gene expression analysis.
Characterize melanin levels using non-invasive skin probes | 1 year
  Obtain average melanin index, fibrosis, and elastimeter values for subjects with dyschromic hypertrophic scar.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Shupp, MD, Principal Investigator — Medstar Health Research Institute
Locations (1):
- MedStar Washington Hospital Center, Washington D.C., District of Columbia, United States

IPD SHARING:
Plan to Share IPD: No